CLINICAL TRIAL: NCT05185284
Title: Open-label Randomized Multicenter Comparative Study on the Efficacy and Safety of AREPLIVIR® (Favipiravir) for Parenteral Administration (PROMOMED RUS LLC, Russia) in Hospitalized Patients With COVID-19
Brief Title: Randomized Multicenter Study on the Efficacy and Safety of Favipiravir for Parenteral Administration Compared to Standard of Care in Hospitalized Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Collaborators: Solyur Pharmaceuticals Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAV-052021
Record Dates: First submitted 2022-01-07; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Areplivir; 2019-nCoV; Favipiravir; Pneumonia; Coronavirus Infections
MeSH Terms: conditions — COVID-19; Pneumonia; Coronavirus Infections | interventions — favipiravir; remdesivir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Areplivir) (Experimental): Arm 1 (n=106) receives the study drug Areplivir for parenteral administration as follows: Day 1 1600 mg 2 times a day, Day 2-10 800 mg 2 times a day. Administration will be done intravenously by drip infusion for 2 hours. The course of treatment is 10 days. The test drug is administered in hospital setting under supervision of a clinical investigator. The test drug is not handed over to the patient.
  Interventions: Drug: Favipiravir
- Standard of care (Active Comparator): Arm 2 (n=108) patients receive standard therapy prescribed in accordance with the recommended treatment regimens included in the Interim Guidelines for the prevention, diagnosis and treatment of new coronavirus infection (COVID-19) approved by the Russian Ministry of Health by decision of the investigator and taking into account the availability of drugs at the study site. Might include Favipiravir tab, Remdesivir or other recommended schemes.
  Standard therapy is administered in hospital setting. Discharge of patients from a hospital is carried out in accordance with the local practice of the study site in compliance with the current sanitary and epidemiological regime.
  Interventions: Drug: Favipiravir; Drug: Remdesivir

INTERVENTIONS:
Drug: Favipiravir — 400 mg, lyophilizate for preparation of concentrate for solution for infusion
  Other Names: Areplivir
  Arms: Favipiravir (Areplivir)
Drug: Favipiravir — 200 mg coated tablets
  Arms: Standard of care
Drug: Remdesivir — 100 mg, lyophilizate for preparation of concentrate for solution for infusion
  Arms: Standard of care

SUMMARY:
This is open-labe randomized multicenter comparative Phase III study conducted in 7 medical facilities. The objective of the study is to assess the efficacy and safety of Favipiravir for parenteral administration compared with the Standard of care (SOC) in hospitalized patients with moderate COVID-19 pneumonia.

DETAILED DESCRIPTION:
Upon signing the informed consent form and screening, 217 eligible patients hospitalized with COVID-19 pneumonia were randomized at a 1:1 ratio to receive either Favipiravir intravenously by drip infusion for 2 hours 1600 mg twice a day (BID) on Day 1 followed by 800 mg BID on Days 2-14 (1600/800 mg), or SOC. The course of treatment by Favipiravir is 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of the Informed Consent Form of the Patient Information Leaflet (PIL) signed and dated by patient.
2. Men and women aged 18 to 80 years inclusive at the time of signing the Informed Consent Form in PIL.
3. Confirmed case of COVID-19 at the time of screening based on SARS-CoV-2 RNA test using nucleic acid amplification (NAA) method. It is acceptable to include a patient with a presumptive COVID-19 diagnosis prior to receiving the results of SARS-CoV-2 RNA test made at the screening stage.
4. Hospital admission due to COVID-19.
5. Moderate severity infection with SARS-CoV-2:

   * Clinical signs:
   * Mandatory: CT pattern typical of a viral lesion (lesion volume is minimal or moderate; CT 1-2).
   * Additional (at least 1 of the following criteria):
   * body temperature > 38 °C;
   * RR > 22/min;
   * shortness of breath on exertion;
   * SpO2 < 95%;
   * Serum CRP > 10 mg/L.
6. Patient's consent to use reliable contraceptive methods throughout the study and within 1 month for women and 3 months for men after its completion. Reliable means of contraception are: sexual abstinence, use of condom in combination with spermicide.

For men (optional): Consent to avoid sexual contact with pregnant women for the duration of the study and for 3 months after its completion.

Women incapable of childbearing may also participate in the study (with past history of: hysterectomy, tubal ligation, infertility, menopause for more than 2 years), as well as men with infertility or a history of vasectomy.

Exclusion Criteria:

1. Hypersensitivity to favipiravir, remdesivir and/or other components of the study drug.
2. Impossibility of CT procedure (for example, gypsum dressing or metal structures in the field of imaging).
3. History of vaccination against COVID-19.
4. History of presumptive or confirmed COVID-19 case of moderate, severe and extremely severe course of the disease.
5. Use of favipiravir or remdesivir within 10 days prior to screening.
6. The need to use drugs from the list of prohibited therapy.
7. Meeting the criteria for severe and extremely severe course of the disease.
8. Need for treatment in the intensive care unit.
9. Impaired liver function (AST and/or ALT ≥ 2 UNL and/or total bilirubin ≥ 1.5 UNL) at the time of screening.
10. Renal impairment (GFR < 60 ml/min) at the time of screening.
11. History of gout.
12. Positive testing for HIV, syphilis, hepatitis B and/or C.
13. Chronic heart failure FC III-IV according to New York Heart Association (NYHA) functional classification (see Appendix 2).
14. Malignancies in the past medical history.
15. Alcohol, pharmacological and/or drug addiction in the past medical history and/or at the time of screening.
16. Schizophrenia, schizoaffective disorder, bipolar disorder, or other history of mental pathology or suspicion of their presence at the time of screening.
17. Severe, decompensated or unstable somatic diseases (any disease or condition that threaten the patient's life or impair the patient's prognosis, and also make it impossible for him/her to participate in the clinical study).
18. Any history data that the investigating physician believes could lead to complication in the interpretation of the study results or create an additional risk to the patient as a result of his/her participation in the study.
19. Patient's unwillingness or inability to comply with procedures of the Study Protocol (in the opinion of physician investigator).
20. Pregnant or nursing women or women planning pregnancy.
21. Participation in another clinical study for 3 months prior to inclusion in the study.
22. Other conditions that, according to the physician investigator, prevent the patient from being included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of Clinical Status Improvement | By Visit 3, approximately 10 days
  Rate of clinical status improvement by WHO categorical ordinal scale of clinical status improvement by 2 or more categories by Day 10. WHO Ordinal Scale for Clinical Improvement (WHO-OSCI), 0 - uninfected (There are no clinical and virological signs of infection), 8 - dead, higher scores mean a worse outcome
Time to Clinical Improvement | 28 days
  Time (in days) to improvement in clinical status by WHO categorical ordinal scale of clinical status improvement

SECONDARY OUTCOMES:
Rate of Clinical Status Improvement | 14 days
  Rate of clinical status improvement by WHO categorical ordinal scale of clinical status improvement by 2 or more categories at Visits 2 (Day 5) and 4 (Day 14)
Rate of Clinical Status Improvement | 14 Days
  Percentage of patients with clinical status of 0 and 1 point according to the WHO categorical ordinal scale of clinical improvement on Days 5, 10 and 14.
End of Fever on Days of study | 14 Days
  Percentage of patients with fever disappearance (body temperature < 37,2 °C in 3 consecutive measurements without antipyretic medication) an Days 5, 10 and 14.
Change in the Level of Lung Damage According to CT | 14 Days
  Assessment of lung injury (degree of damage by "empirical" visual scale and % of patients) according to CT data comparing to baseline. The number of patients in whom by the end of therapy there was an improvement in the condition of the lungs (a decrease in the volume of the lesion according to CT)
Rate of Viral Elimination | 14 days
  Percentage of patients with SARS-CoV-2 elimination (negative test for SARS-CoV-2 by NAA method) on Days 5, 10, and 14.
Rate of Transfer to the Intensive Care Unit | 28 days
  Percentage of patients transferred to intensive care unit
Rate of the Use of Non-invasive Lung Ventilation | 28 Days
  Percentage of cases with non-invasive lung ventilation
Rate of the Use of Mechanical Ventilation | 28 Days
  Percentage of cases with mechanical lung ventilation (% of patients)
Mortality | 28 Days
  Incidence of fatal cases (% of patients)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Pushkar, MD, Academic, Principal Investigator — Moscow State Clinical Hospital №50
Locations (6):
- Russia (6):
  - Regional budgetary health care institution "Ivanovo Clinical Hospital named after Kuvaevs", Ivanovo
  - State Budgetary Institution of Healthcare of the City of Moscow "City Clinical Hospital No. 24 of the Department of Healthcare of the City of Moscow", Moscow
  - State Clinical Hospital №50, Moscow
  - Regional Clinic Hospital of Ryazan, Ryazan
  - Medical institute Ogarev Mordovia State university, Saransk
  - Smolensk clinical hospital №1, Smolensk

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: January 2022